CLINICAL TRIAL: NCT02800889
Title: A Phase 1, Dose-Escalation Study of Pixantrone Monotherapy in Pediatric Patients With Relapsed or Refractory Cancer
Brief Title: Dose-Escalation Study of Pixantrone Monotherapy in Pediatric Patients With Relapsed or Refractory Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn; no participants enrolled
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIX111
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma; Solid Tumor (Excluding CNS)
Keywords: relapsed; refractory; solid tumors
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — pixantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: Pixantrone (Experimental): Each patient will receive pixantrone monotherapy administered intravenously once on days 1, 8, and 15 up to six 28-day cycles of pixantrone monotherapy, with two additional cycles in patients who continue to benefit from treatment. At least 6 patients each from Age Cohorts 1 and 2 will be accrued into dose escalation cohorts. The study will be opened to patients of Age Cohort 3 only after at least 6 patients in Age Cohorts 1 and 2 (combined) have been evaluated for toxicity. During the dose escalation phase, participants who are inevaluable for DLT for reasons unequivocally unrelated to toxicity will be replaced. Expansion cohort accrual quota-At least 15 evaluable patients treated with the MTD/optimal dose will be accrued in total, of which 7 patients will be in Age Cohort 2.
  Interventions: Drug: Pixantrone

INTERVENTIONS:
Drug: Pixantrone — Pixantrone
  Other Names: Pixantrone (BBR 2778)

SUMMARY:
This is a phase 1, open-label, dose escalation study to evaluate the safety, pharmacokinetics, and antitumor activity of pixantrone in pediatric patients with relapsed or refractory solid tumors (excluding those with CNS tumors) or lymphoma.

DETAILED DESCRIPTION:
Approximately thirty-five eligible patients will receive up to six 28-day cycles of pixantrone monotherapy, with two additional cycles in patients who continue to benefit from treatment. Each patient will receive pixantrone administered intravenously on days 1, 8, and 15 of each 28-day cycle. There will be three age cohorts, defined as age cohort 1 (12 to less than 18 years, plus young adults (ages 18-21 years)), age cohort 2 (5 to less than 12 years), and age cohort 3 (6 months to less than 5 years). During dose escalation, three patients will first be accrued to the starting dose level. If no DLTs are identified, that dose level will be declared to not exceed the MTD and three patients will be accrued to the next higher dose level. Each subsequent dose-escalation level will be accrued per the DLT/MTD determination schema above. Planned sequential dose-escalation phase will receive 40 mg/m2, 50 mg/m2, 60 mg/m2 or 70 mg/m2 of pixantrone base (on days 1, 8 and 15), as tolerated, based on DLT evaluation.Dose escalations will follow a standard 3+3 patient cohort escalation plan. No patients from Age Cohort 3 will be enrolled until 6 patients from age cohorts 1 and 2 (combined) are evaluable for toxicity. After the MTD has been determined, an expansion phase will be accrued in order to gain better estimates of the safety, tolerability, and anti-tumor activity of pixantrone monotherapy in pediatric patients when treated at the MTD. Patients will be offered 3 years of post-study extension phase follow-up with periodic assessments of cardiac function parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or guardian have signed an Informed Consent Form and Assent approved by the Institutional Review Board or Institutional Ethics Committee, as appropriate and necessary, on a per-age basis
2. Age 6 months to 21 years old (initial qualifying diagnosis must have been made at or before the age of 18 and the patient must be under the care of a pediatric hematologist/oncologist)
3. Patient received a diagnosis of lymphoma or any non-hematologic malignancy (except central nervous system [CNS] tumors) for which the patient is considered relapsed or refractory. (NOTE: CNS metastases are allowable in patients who are deemed not at risk for progression during the first 30 days, who are neurologically stable, and, if on corticosteroids, have been on a stable corticosteroid dose for at least 2 weeks.) Patients who have >1 malignancy ongoing during screening are not eligible
4. Patient must have one or more of the following treatment statuses:

   * Has failed at least 2 prior lines of chemotherapy
   * Has no curative chemotherapy treatment option available
   * Is not considered a candidate for available chemotherapy treatment options
5. In dose-escalation accrual, patients may have un-measurable disease (such as bone marrow/bone involvement or diffuse tumors)
6. In dose-escalation accrual, patients may have un-measurable disease in cases where the standard of care would indicate the need for adjuvant chemotherapy after definitive surgery or radiation, but for whom no standard chemotherapy options are available
7. In expansion cohort accrual, patients must have disease that is evaluable or measurable for response and progression per standard criteria for their diagnosis (Refer to the Appendices: RECIST 1.1 Criteria for Evaluation of Solid Tumors, Including Neuroblastoma, Appendix 18.4], Evaluation of Neuroblastoma [Appendix 18.6], and the Lymphoma Staging and Disease Response Criteria [Appendix 18.5])
8. Karnofsky-Lansky performance status (as per age of patient) ≥50 (Appendix 18.1)
9. Patient must have one or more of the following cardiac function measurements by echocardiogram:

   * Left ventricular ejection fraction (LVEF) ≥55%
   * Left ventricular shortening fraction (LVSF) ≥27%
10. Hemoglobin ≥8 g/dL (can be post-transfusion)
11. Platelet count ≥75 × 109/L
12. Absolute neutrophil count (ANC) ≥0.75 × 109/L
13. Serum direct/conjugated bilirubin ≤1.5 × upper limit of normal (ULN); patients with clinically diagnosed Gilbert's syndrome and total bilirubin ≤5 × ULN may be enrolled
14. Aspartate aminotransferase (AST; also called serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT; also called serum glutamic-pyruvic transaminase [SGPT]) ≤2.5 × ULN, or ≤5 × ULN if elevation is due to hepatic involvement by tumor
15. Serum creatinine ≤2 × ULN
16. Patients must meet the following criteria with respect to prior cancer therapy, radiotherapy, and stem cell transplants:

    1. Myelosuppressive chemotherapy: At least 3 weeks must have elapsed since the completion of myelosuppressive chemotherapy (4 weeks if prior nitrosourea) and resolution of all nonhematologic toxicities to ≤grade 1.
    2. Biologic (anti-neoplastic agent):

       * Oral tyrosine kinase inhibitors or other similar agents. At least 7 days must have elapsed since the completion of therapy with a biologic agent and all non-hematologic toxicities must have resolved to ≤grade 1 prior to enrollment
       * Anti-IGFR-1R and other monoclonal antibodies: the shorter of 3 half-lives or 6 weeks must have elapsed since previous monoclonal antibody therapy and resolution of all non-hematologic toxicities to ≤grade 1 prior to enrollment
    3. Myeloid Growth Factor: Must not have received within 1 week prior to entry into this study (2 weeks in the case of PEG-filgrastim)
    4. Radiotherapy: At least 4 weeks must have elapsed and all non-hematologic toxicities must have resolved to ≤grade 1 prior to enrollment. Previously radiated lesions cannot be used to assess response unless those sites are the sites of disease progression
    5. Stem cell transplant (SCT): For autologous SCT, ≥3 months must have elapsed. For allogeneic SCT, ≥6 months must have elapsed and there must be no evidence of active graft versus host disease
17. All acute toxicities related to prior treatment recovered to grade ≤1 , except alopecia and hematologic parameters specified in the inclusion criteria
18. Willingness and ability to comply with the visit schedule and assessments required by the study protocol, including effective birth control (Section 5.4) for sexually active patients

Exclusion Criteria:

1. Investigator-predicted life expectancy of less than two months
2. Investigator-predicted inability to tolerate pixantrone monotherapy treatment adverse effects for less than two months
3. Prior anthracycline treatment with a cumulative dose exceeding 450 mg/m2 (calculated based on doxorubicin equivalents)
4. Active National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) ≥grade 3 infection, or a lower grade infection deemed resistant or refractory to available antimicrobial agents, or infection requiring ongoing antibiotic treatment
5. Major surgery ≤7 days and/or with incomplete/inadequate wound healing prior to start of study treatment
6. Known acute or chronic hepatitis B or hepatitis C virus infection
7. Known seropositivity for human immunodeficiency virus (HIV)
8. Any experimental/investigational therapy ≤28 days prior to start of study treatment
9. Myocardial infarction within the past 6 months
10. New York Heart Association class II, III or IV heart failure
11. Any contraindication, known allergy, or hypersensitivity to any investigational drug(s)
12. Pregnant or lactating
13. Planned radiotherapy or surgical procedures for the qualifying malignancy
14. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study procedures or follow-up schedules
15. Other severe and/or uncontrolled medical disease that could compromise participation in the study, or any medical or psychiatric condition that, in the opinion of the investigator, would make study drug administration hazardous or obscure the interpretation of data

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose level at which no more than 1/6 patients experience DLT | 28 days
  Dose Escalation- The study will follow a standard 3+3 patient cohort escalation design, evaluating up to 4 dose levels.
Anti-tumor activity of pixantrone at the MTD | approx. 1 year
  Dose Expansion Cohort- Anti-tumor activity will be summarized by disease type, dose level, and age cohort for all patients in the evaluable population. The best overall response rate, defined as the proportion of patients that achieved a complete or partial response, will be summarized by disease type and a 95% confidence interval will be provided. A similar summary will be provided for the complete response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Mascarenhas, MD. MS., Principal Investigator — CHLA
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States